CLINICAL TRIAL: NCT01142986
Title: Evaluating Three Methods for Helping Syringe Exchangers Begin Methadone Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2R01DA012347 (NIH)
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Substance Abuse Disorder
Keywords: Methadone; Syringe exchange; Treatment retention; Voucher incentives
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Threshold Stepped Care (LTSC) (Experimental): Subjects in this condition will receive low intensity care during the first 3-months (13 weeks) of study participation, and usual counseling care during the final 3-months (13 weeks) of participation.
  Interventions: Behavioral: Low intensity care
- Voucher-Based Stepped Care (VBSC) (Experimental): Subjects in this condition will receive usual counseling care during the entire 6 months of study participation. They will receive voucher reinforcement, and will have the opportunity to earn voucher incentives during the first 3-months of care (13 weeks).
  Interventions: Behavioral: Voucher reinforcement
- Routine Stepped-Care (RSC) (No Intervention): Subjects in this condition will receive usual counseling care during the entire 6-month study (26 weeks).

INTERVENTIONS:
Behavioral: Low intensity care — During the first 3-months (13 weeks), subjects will be scheduled to attend one individual counseling session per month. Subjects will not be required to attend any group counseling sessions during this time. After the first 3-months of care, subjects will start usual counseling care, at which time they will be required to attend one individual counseling session per week, and may be required to attend additional individual and group counseling sessions each week for missed sessions or continued use of drugs or alcohol.
  Arms: Low Threshold Stepped Care (LTSC)
Behavioral: Voucher reinforcement — Subjects will receive usual counseling care during the 26 weeks of study participation.They will be required to attend one individual counseling session per week, and will be required to attend additional individual and group sessions each week for missed session or continued use of drugs or alcohol.In addition, subjects in this condition will have the opportunity to earn voucher incentives each week during the first 13 weeks of care.These incentives can be earned by taking daily methadone doses and attending all scheduled counseling sessions (individual and group).The first voucher is worth $12.00, and each voucher after that is worth an additional $13.50. Bonuses of $30.00 will be awarded for each 3 consecutive weeks of compliance.The total amount possible to earn in the study is $1329.00. Each week that the subject is not compliant,they will not earn a voucher and the value of the next voucher will be reset to $12.00.The vouchers can be used for goods and services in the community.
  Arms: Voucher-Based Stepped Care (VBSC)

SUMMARY:
This research is being done to evaluate the effectiveness of three different treatment strategies for helping subjects begin and adjust to methadone maintenance treatment at Addiction Treatment Services (ATS). Subjects will be randomly assigned to one of three treatment conditions: 1) Voucher-Based Stepped Care (VBSC) induction, 2) Low-threshold Stepped Care (LTSC) induction, or 3) Routine Stepped Care (RSC) induction. It is hypothesized that subjects in both the VBSC and LTSC condition will remain in treatment longer than subjects in the RSC condition. In addition, it is hypothesized that VBSC and LTSC subjects will have less drug-positive urine samples and will report less infectious disease risk behaviors than RSC subjects.

DETAILED DESCRIPTION:
This study will evaluate two alternative methods of inducting syringe exchange referrals into routine methadone treatment. The sample (N=390) will be opioid-dependent injection drug users referred by the Baltimore Needle Exchange Program (BNEP) for routine outpatient methadone treatment using a stepped care model. Subjects will be randomly assigned to one of three 3-month treatment induction conditions: 1) Low Threshold Stepped Care induction (LTSC), 2) Voucher-Based Stepped Care induction (VBSC), or 3) Routine Stepped-Care induction (RSC). The LTSC condition will noticeably reduce treatment demands on new admissions during the 90-day induction period and is conceptually related to an interim maintenance schedule. It is expected to increase patient recognition of the reinforcing effects and benefits of methadone, improve the transition to more comprehensive schedules of care, and increase early retention. The VBSC condition adds an attendance reinforcement intervention to the routine stepped care induction schedule over the first 90-days of treatment. It is expected to improve early treatment engagement and retention. Subjects in each of these conditions will transition to routine stepped-care (no voucher-based reinforcement) following the 90-day induction period. The RSC condition will serve as a comparison group and represents routine care in the program where the study will be conducted. All subjects will be followed for 6-months. Retention, drug use (via urinalysis and self-report), and other infectious disease risk behaviors (e.g., syringe sharing; number of injections) are the primary outcome measures. The proposed design will also test mediational models to evaluate changes in objective indices of engagement (methadone and counseling adherence) and psychological constructs (treatment readiness and satisfaction) as predictors of outcome. Regression models will be used to evaluate the amount of reduction of drug use necessary to effect varying amounts of change in HIV risk behavior. Finally, data will be collected and compared on the treatment costs of each induction strategy.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Baltimore Needle Exchange Program (BNEP)
* Expressed interest in treatment with methadone.

Exclusion Criteria:

* Pregnancy
* Currently in a treatment program using methadone or other agonist medications
* Failure to meet DSM-IV criteria for opioid physical dependence and CSAT guidelines for long-term use of opioid agonist medications
* Presence of an acute medical problem that requires immediate and intense medical management (e.g., AIDS defining illness; tuberculosis; unstable diabetes, hypertension, and other problems)
* Presence of a formal thought disorder, delusions, hallucinations, or imminent risk of harm to self or others (symptoms commonly associated with schizophrenia, bipolar disorder, and other major mental illnesses).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Treatment retention and time to dropout | Weekly for 26 weeks
  The length of time subjects remain in treatment is tracked throughout the study. Retention will be assessed as: 1) percent of subjects remaining in treatment at 3 and 6-months, and 2) time to dropout.
Substance use | Weekly for 26 weeks
  Subjects are required to leave weekly urine specimens (for 12-weeks) which are tested for drugs of abuse. Percent positive for opiates, cocaine, benzodiazepines, and cannabis will be evaluated weekly. Self-report use will be assessed for subjects in and out of treatment.
Infectious disease risk behaviors | Monthly for 6 months
  Risk behavior will be assessed via the the Risk Assessment Battery (RAB) and Addiction Severity Index at baseline and monthly intervals throughout the study for subjects in and out of treatment.

SECONDARY OUTCOMES:
Other problem severity | Monthly for 6 months
  Addiction Severity Index (ASI) composite scores will be assessed at baseline and at monthly intervals.
Counseling engagement | Weekly for 26 weeks
  Total number of individual and group counseling sessions attended, as well as adherence to scheduled sessions (i.e. attended/scheduled), will be monitored.
Methadone dose | Weekly for 26 weeks
  Mean methadone dose, days receiving methadone, and dose adequacy will be evaluated.
Treatment readiness | Monthly for 6 months
  Treatment readiness will be assessed via the TCU Treatment Motivation Scales (TMS) at baseline and monthly intervals.
Treatment satisfaction | Monthly for 6 months
  The Client Satisfaction Questionnaire (CSQ) will assess treatment satisfaction at baseline and monthly intervals.
Use of syringe exchange and other community-based services | Monthly for 6 months
  Days of syringe exchange program (SEP) use, number of syringes exchanged, and use of other community-based medical and psychosocial resources (e.g. emergency room, psychiatric and other treatment facilities, shelters, hospitalization) will be assessed for participants in and out of treatment at baseline and monthly intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kidorf, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services, Baltimore, Maryland, United States